CLINICAL TRIAL: NCT02253628
Title: The Acute Effect of Coffee Consumption on Salivary Gastrin, Alpha-amylase and Cortisol Concentrations, on Self-reported Gastrointestinal Symptoms, on Self-reported Psychometric Assessments and on Blood Pressure.
Brief Title: The Acute Effect of Coffee Consumption on Stomach, Self-reported Gastrointestinal Symptoms and Stress.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Lecturer of Nutrition and Metabolism, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 340302
Record Dates: First submitted 2014-09-19; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Stress; Signs and Symptoms, Digestive; Blood Pressure; Increased Secretion of Gastrin
Keywords: Coffee; Gastrin; Alpha-amylase; Cortisol; Self-reported gastrointestinal symptoms; Self-reported stress; Blood pressure
MeSH Terms: conditions — Signs and Symptoms, Digestive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Trial 1 (Experimental): Forty healthy men and women, with normal body weight. Volunteers consumed randomly 4 coffee beverages with 160 mg caffeine (hot instant coffee, cold instant coffee, cold espresso, hot filter coffee).
  Interventions: Other: Cold espresso; Other: Hot instant coffee; Other: Cold instant coffee; Other: Hot filter coffee
- Trial 2 (Experimental): Forty healthy men and women, with normal body weight. Volunteers consumed randomly 4 coffee beverages with 160 mg caffeine (hot instant coffee, cold instant coffee, cold espresso, hot filter coffee).
  Interventions: Other: Cold espresso; Other: Hot instant coffee; Other: Cold instant coffee; Other: Hot filter coffee
- Trial 3 (Experimental): Forty healthy men and women, with normal body weight. Volunteers consumed randomly 4 coffee beverages with 160 mg caffeine (hot instant coffee, cold instant coffee, cold espresso, hot filter coffee).
  Interventions: Other: Cold espresso; Other: Hot instant coffee; Other: Cold instant coffee; Other: Hot filter coffee
- Trial 4 (Experimental): Forty healthy men and women, with normal body weight. Volunteers consumed randomly 4 coffee beverages with 160 mg caffeine (hot instant coffee, cold instant coffee, cold espresso, hot filter coffee).
  Interventions: Other: Cold espresso; Other: Hot instant coffee; Other: Cold instant coffee; Other: Hot filter coffee

INTERVENTIONS:
Other: Cold espresso — Volunteers consumed cold espresso with 160 mg caffeine. Salivary gastrin, alpha-amylase and cortisol and self-reported GI symptoms and stress were collected at fasting and postprandially.
  Other Names: Buondi prestige
Other: Hot instant coffee — Volunteers consumed hot instant coffee with 160 mg caffeine. Salivary gastrin, alpha-amylase and cortisol and self-reported GI symptoms and stress were collected at fasting and postprandially.
  Other Names: Nescafé Classic
Other: Cold instant coffee — Volunteers consumed cold instant coffee with 160 mg caffeine. Salivary gastrin, alpha-amylase and cortisol and self-reported GI symptoms and stress were collected at fasting and postprandially.
  Other Names: Nescafé Classic
Other: Hot filter coffee — Volunteers consumed hot filter coffee with 160 mg caffeine. Salivary gastrin, alpha-amylase and cortisol and self-reported GI symptoms and stress were collected at fasting and postprandially.
  Other Names: Nestlé Professional Plantage Filter Coffee

SUMMARY:
This study investigated the acute effect of the consumption of four different kinds of coffee (hot and cold instant coffee, cold espresso and hot filter coffee) with the same caffeine content on salivary gastrin, cortisol and alpha-amylase concentrations, on self-reported gastrointestinal symptoms and on psychometric assessments in healthy individuals.

DETAILED DESCRIPTION:
Coffee consumption is very common in Greece. Many of the consumers support that certain types of coffee and especially instant coffee cause gastrointestinal symptoms in healthy individuals. Up to now, few studies have investigated the relationship between coffee consumption, gastrointestinal symptoms and stress in healthy individuals with conflicting results.Coffee consumption is related with increased gastric acid and gastrin secretion, however it does not seem to affect stomach or stomach walls. Stress, which characterizes modern lifestyle, also is found to increase gastric acid and gastrin secretion and seems to be exclusively responsible for gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Stable body weight for at least 1 month prior to study enrollment.

Exclusion Criteria:

* If one volunteer consumed breakfast more than three days a week, their daily caffeine intake was over 500 mg caffeine, was taking medication, their psychological state was strongly influenced by some exogenous factor (e.g. moving to a new house, new job, divorce e.t.c.), was on hypocaloric diet for weight loss, was smoking more than five cigarettes a day, was an athlete with very vigorous physical activity (> 4 hours vigorous exercise a day), had a history of gastrointestinal disorders (e.g. gastroesophageal reflux disease (GERD), irritable bowel syndrome, diarrhea, ulcers e.t.c.), depression, diabetes, kidney disease, hypertension, blood disorders, liver disease, unregulated hyper - or hypothyroidism, arrhythmia, heart disease, cancer, vascular disease, recent surgery, or severe psychiatric disorders was automatically excluded from the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Salivary gastrin and self-reported gastrointestinal symptoms | 4 weeks
  The volunteers visited the lab after an 8-hour fasting. Saliva samples were taken at fasting for the determination of fasting salivary gastrin. After the consumption of coffee, saliva samples were taken at 15, 30, 60' for the determination of gastrin. Saliva samples were collected by the method "Salivette". Saliva was carried out by chewing a swab for about 1 minute. Then, the swab was returned to the Salivette and the container was centrifuged and saliva sample was obtained. The samples were stored at - 20 degrees of Celsius. Gastrin was determined by an immunoenzymatic method. In order to record the effects of coffee consumption on gastrointestinal symptoms, the participants completed a visual analogue scale every time saliva samples were collected (time 0', 15', 30', 60', 120', 180'). The visual analogue scale (1 = not at all to 10 = very) included 12 questions about gastrointestinal symptoms.

SECONDARY OUTCOMES:
Blood pressure, energy intake and physical activity | 4 weeks
  The aim was to investigate if blood pressure, energy intake and physical activity changed during the intervention. Blood pressure was measured three times in a sitting position after 15 minutes of rest by a mercury sphygmomanometer at the beginning and ending of each trial respectively. There was a 2-minute interval between measurements. Then, the average blood pressure measurements were calculated. Dietary intake was analyzed by Diet Analysis Plus (version 6.1). The database was extensively modified to include new foods and recipes. Physical activity was estimated by using metabolic equivalents of different activities performed by the volunteers the previous 7 days. Then, mean daily energy expenditure was estimated.
Salivary cortisol and alpha-amylase | 4 weeks
  The volunteers visited the lab after an 8-hour fasting. Saliva samples were taken at fasting for the determination of fasting salivary cortisol and alpha-amylase. After the consumption of coffee, saliva samples were taken at 15, 30, 60' for the determination of alpha-amylase and at 60, 120, 180' for cortisol determination.Saliva samples were collected by the method "Salivette". Saliva was carried out by chewing a swab for about 1 minute. Then, the swab was returned to the Salivette and the container was centrifuged and saliva sample was obtained. The samples were stored at - 20 degrees of Celsius. Cortisol was determined by an immunoenzymatic method. Alpha-amylase was determined by a kinetic enzyme assay kit.
Self-reported sentiments, mood and stress. | 4 weeks
  In order to record the effects of coffee consumption on stress and on sentiments and mood the participants completed the Zung self-assessment anxiety scale and a visual analogue scale every time saliva samples were collected (time 0', 15', 30', 60', 120', 180'). The Zung self-assessment anxiety scale included 20 questions, which were designed to assess how the volunteers felt the moment completing the questionnaire. The visual analogue scale (1 = not at all to 10 = very) included 17 questions about stress, sentiments and mood.

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens

REFERENCES:
- [Derived] Papakonstantinou E, Kechribari I, Sotirakoglou Kappa, Tarantilis P, Gourdomichali T, Michas G, Kravvariti V, Voumvourakis K, Zampelas A. Acute effects of coffee consumption on self-reported gastrointestinal symptoms, blood pressure and stress indices in healthy individuals. Nutr J. 2016 Mar 15;15:26. doi: 10.1186/s12937-016-0146-0. PMID 26979712